CLINICAL TRIAL: NCT07207447
Title: Validity of the Non-union Scoring System in Management of Long Bone Fracture Non-union: A Prospective Study
Brief Title: Validity of the Non-union Scoring System in Management of Long Bone Fracture Non-union
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FMASU MD21/2022
Record Dates: First submitted 2025-09-12; First posted 2025-10-06 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Fracture Non Union
Keywords: NUSS; Non-union Scoring System; Fracture Non-Union; Bone defect
MeSH Terms: conditions — Fractures, Ununited | interventions — Amputation, Surgical

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- NUSS group 1 (Active Comparator)
  Interventions: Procedure: Improving the stability and re-fixation with different modalities
- NUSS group 2 (Active Comparator)
  Interventions: Procedure: Re-fixation with biological stimulation
- NUSS group 3 (Active Comparator)
  Interventions: Procedure: complex care with non-union resection and bone reconstruction
- NUSS group 4 (Active Comparator)
  Interventions: Procedure: Amputation

INTERVENTIONS:
Procedure: Improving the stability and re-fixation with different modalities — Improving the stability and re-fixation with different modalities such as exchange plate with longer plate, intramedullary nailing, exchange nailing with larger diameter, plating over nail or dynamization of intramedullary nail.
  Arms: NUSS group 1
Procedure: Re-fixation with biological stimulation — Re-fixation with biological stimulation such as bone grafting, either with plate and bone graft, plate over nail and graft, or with external fixation with LRS or Ilizarov and grafting in one stage or two stages.
  Arms: NUSS group 2
Procedure: complex care with non-union resection and bone reconstruction — complex care with non-union resection and bone reconstruction, including resection of the non-union and dealing with the defect with bone transport, either direct transport or staged with cement spacer and later bone transport, Masquelet technique or acute compression and lengthening with another osteotomy.
  Arms: NUSS group 3
Procedure: Amputation — Amputation with consideration of prosthesis.
  Arms: NUSS group 4

SUMMARY:
The aim of this study is to apply Calori Non union Scoring System on long bone non-union cases and evaluate the results of treatment o f the patients according to the score.

DETAILED DESCRIPTION:
The aim of this study is to apply Calori Non union Scoring System on long bone non-union cases and evaluate the results of treatment o f the patients according to the score. The study will be on patients with lower limb long bone diaphyseal fracture non-union. All patients will be assessed preoperatively by Clinical Evaluation: History, general examination, local examination, radiological evaluation: Plain X-ray films showing joint above and joint below the non-union site, laboratory Investigations: CBC, ESR, CRP and HbA1c. For patient allocation, patients will be divided into four groups according to the NUSS score, with group one (0-25 points) who underwent improving the stability and re-fixation with different modalities such as exchange plate with longer plate, intramedullary nailing, exchange nailing with larger diameter, plating over nail or dynamization of intramedullary nail. Group two (26-50 points) underwent re-fixation in addition to biological stimulation such as bone grafting, either with plate and bone graft, plate over nail and graft, or with external fixation with LRS or Ilizarov and grafting in one stage or two stages. Group three (51-75 points) required more complex care with resection of the non-union and dealing with the defect with bone transport, either direct transport or staged with cement spacer and later bone transport, Masquelet technique or acute compression and lengthening with another osteotomy. Group four (76-100 points) underwent amputation with consideration of prosthesis. The patients will be followed up at regular intervals as regard radiological and clinical evaluation until full union is achieved or non-union is established. The assessment includes; clinical and functional assessment based on pain at the fracture site and recovery of the usual activities or work, and radiological assessment based on plain radiograph x-rays, CT scan if needed to assess union. Radiological union is considered based on the presence of bridging callus (3/4 of cortices) in both anteroposterior and lateral views.

ELIGIBILITY:
Inclusion Criteria:

* Sex: both sexes.
* Age: Above 18 years old.
* Lesion: Tibial or femoral bone non-union.

Exclusion Criteria:

* Skeletal immaturity.
* Any immunosuppressive drug therapy.
* Autoimmune disease.
* Neoplasia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-02-10 (Actual); Primary Completion 2024-07-10 (Actual); Study Completion 2024-08-10 (Actual)

PRIMARY OUTCOMES:
Radiological Fracture Union | According to each group ranging from 5 months in group 1, 7 in group 2 and up to 12 months in group 3
  Radiological fracture union is considered based on the presence of bridging callus (3/4 of cortices) in both anteroposterior and lateral views in x rays.
Clinical Fracture Union | According to each group ranging from 4 months in group 1, 6 in group 2 and up to 11 months in group 3.
  Clinical fracture union assessment is based on presence or absence of pain at the fracture site.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Abbasia, Egypt